CLINICAL TRIAL: NCT01463527
Title: Using Capnography to Reduce the Incidence of Hypoxia in Children During Moderate Sedation in the Pediatric Emergency Department: A Randomized Controlled Trial
Brief Title: Using Capnography to Reduce Hypoxia During Pediatric Sedation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 0904005003
Record Dates: First submitted 2011-10-24; First posted 2011-11-02 (Estimated); Results first posted 2014-08-04 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2017-12

CONDITIONS: Hypoventilation; Hypoxia
Keywords: Hypoventilation during sedation; Hypoxia associated with hypoventilation
MeSH Terms: conditions — Hypoventilation; Hypoxia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Open Capnography (Experimental)
  Interventions: Device: Nellcor NPB-70 Capnograph
- Capnography Blind (Placebo Comparator)
  Interventions: Device: Nellcor NPB-70 Capnograph

INTERVENTIONS:
Device: Nellcor NPB-70 Capnograph — Use of capnography as an additional monitor during sedation to detect hypoventilation and apnea prior to declines in pulse oximetry and clinical examination findings

SUMMARY:
The investigators hypothesize that the addition of capnography during moderate sedation will improve recognition of hypoventilation and apnea. This will lead to an increased frequency of staff interventions such as verbal or physical stimulation for these events in order to improve ventilation which will in turn lead to a reduction in the frequency of oxygen desaturations. If capnography proves to be effective in creating earlier detection and intervention for hypoventilation and apnea during moderate sedation provided by non-anesthesiologists, this device can be used in a variety of clinical settings to enhance patient safety.

ELIGIBILITY:
Inclusion Criteria:

* Children 1-20 years old who require IV sedation in the Pediatric Emergency Department at Yale-New Haven Children's Hospital

Exclusion Criteria:

* Unable to tolerate nasal-oral cannula
* Conditions that effect end-tidal carbon dioxide measurement (active asthma, diabetic ketoacidosis, severe dehydration or trauma)
* Intubation

Ages: 1 Year to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 167 (Actual)
Dates: Start 2011-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Langhan, MD, Principal Investigator — Yale University
Locations (1):
- Yale-New Haven Children's Hospital, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Langhan ML, Shabanova V, Li FY, Bernstein SL, Shapiro ED. A randomized controlled trial of capnography during sedation in a pediatric emergency setting. Am J Emerg Med. 2015 Jan;33(1):25-30. doi: 10.1016/j.ajem.2014.09.050. Epub 2014 Oct 5. PMID 25445871

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Capnography: Staff members able to view capnography monitor during sedation.
- Capnography Blind: Staff members blinded to capnography screen and alarms turned off during sedation.
Period: Overall Study
Arm/Group | Open Capnography | Capnography Blind
Started | 83 | 84
Completed | 77 | 77
Not Completed | 6 | 7
Not completed — Protocol Violation | 1 | 1
Not completed — Crying >20% of sedation | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Capnography Blind: Staff members were blinded to screen on capnography monitor and all alarms turned off for the sedation.
- Total: Total of all reporting groups
Arm/Group | Open Capnography | Capnography Blind | Total
Number analyzed (Participants) | 77 | 77 | 154
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.6 (5.1) | 8.2 (4.8) | 8.4 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 34 | 65
  Male | 46 | 43 | 89
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 13 | 26
  White | 59 | 60 | 119
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 4 | 9
Indication for sedation [Number; unit: participants]
  Fracture reduction | 43 | 42 | 85
  Laceration repair | 13 | 16 | 29
  Incision and drainage of abscess | 16 | 12 | 28
  Arthorcentesis | 2 | 3 | 5
  Dislocation | 1 | 4 | 5
  Other | 2 | 0 | 2
Weight [Mean (Standard Deviation); unit: kg] | 35.8 (20.8) | 35.8 (21.8) | 35.8 (21.3)

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Staff Interventions for Hypoventilation.
Description: These include verbal or physical stimulation, administration of supplemental oxygen, bag-valve mask ventilation, or use invasive airway devices.
Time Frame: Every 30 seconds during sedation; this is on average 30 minutes (range 10-240 minutes)
Measure: Mean (Full Range); unit: Events per patient minute of sedation
Groups:
- Open Capnography: Staff able to view capnography monitor during sedation.
- Capnography Blind: Staff blinded to capnography screen and alarms turned off during sedation.
Arm/Group | Open Capnography | Capnography Blind
Number analyzed (Participants) | 77 | 77
Events per patient minute of sedation | 0.39 [0 to 2.084] | 0.396 [0 to 2.030]
Statistical Analysis 1: Comparison: Open Capnography vs Capnography Blind; Odds of intervention in capnography open group as compared to capnography blind group after adjusting of age and length of sedation; Test type: Superiority or Other; Odds Ratio (OR) = 0.31, 95% CI 2-sided [0.17 to 0.57]

2. Secondary Outcome: Frequency of Hypoxia Defined as Pulse Oximetry Less Than 95%.
Description: While there were 77 patients per group, each patient had vital signs measured every 30 seconds for the duration of their stay. This resulted in a variable amount of time points (data points) recorded per patient. Our event frequency was the number of events (outcome measure of abnormal vital signs) per number of time points for each patient. This is presented as an event rate.
Time Frame: Every 30 seconds during sedation; this is on average 30 minutes (range 10-240 minutes)
Measure: Mean (Full Range); unit: rate of total events/total time points
Units Other Than Participants: Total Number of Time Points per Group
Arm/Group | Open Capnography | Capnography Blind
Number analyzed (Participants) | 77 | 77
Number analyzed (Total Number of Time Points per Group) | 4330 | 4264
rate of total events/total time points | 0.024 [0.000 to 0.400] | 0.016 [0.000 to 0.176]
Statistical Analysis 1: Comparison: Open Capnography vs Capnography Blind; Test type: Superiority; p = 0.30, GEE (Generalized Estimating Equation)

ADVERSE EVENTS:
Time Frame: During time of sedation in emergency department, an average of 36 minutes
Description: No serious adverse events were recorded.
Arm/Group | Open Capnography | Capnography Blind
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/77
Other Adverse Events (participants affected / at risk) | 0/77 | 0/77

LIMITATIONS AND CAVEATS:
No serious adverse events were recorded. Since these events are rare and this study was not powered to detect them, we are unable to predict how capnography may have impacted staff behavior and patient outcomes for these less frequent events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No